CLINICAL TRIAL: NCT04853004
Title: Studies of Ongoing and Completed SARS-CoV-2 Infection (Which Causes COVID-19) Within the Healthcare in Stockholm County, With Regard to Vaccinations.
Brief Title: Current and Past SARS-CoV-2 Infection and COVID-19 in Healthcare With Regard to Vaccinations
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Joakim Dillner, MD, PhD, Karolinska Institutet
Other Study IDs: Covid19_7
Record Dates: First submitted 2021-04-19; First posted 2021-04-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: SARS-CoV 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Personnel in health and care in Stockholm County, who have previously participated in a study where data on sick leave, SARS-Cov2 infections and SARS-CoV2 antibody levels were collected and documented form the study cohort.
  Interventions: Diagnostic Test: SARS-CoV2 antibody measurement

INTERVENTIONS:
Diagnostic Test: SARS-CoV2 antibody measurement — Blood samples for serology, collected immediately prior to and five to ten weeks after vaccination against SARS-CoV2, to be analyzed for the presence of SARS-CoV-2 antibodies.

SUMMARY:
To investigate the incidence of SARS-CoV-2 infections after vaccination, to monitor the development of SARS-CoV-2 antibody levels after vaccination and to compare this in relation to both previous health & disease, previous antibody responses and in relation to future disease occurring after vaccination.

DETAILED DESCRIPTION:
The purpose of the study is to analyze the effect of and possible side effects of SARS-CoV2 vaccinations in the cohort study where data on sick leave, SARS-Cov2 infections and SARS-CoV2 antibody levels are well documented even before vaccination.

The main outcome measures are the presence of SARS-CoV-2 (ongoing infection) and the presence of antibodies to SARS-CoV-2.

For the vaccination effect, the factors that are primarily associated with protection against infection are analyzed, such as age, sex, workplace, antibody response to SARS-CoV-2 and vaccination date.

The analyzes are planned to be performed with multivariate logistic regression with Relative Risk as the outcome measure.

Data from the analysis of virus antibodies are planned to be performed divided into whether low, medium or high levels of antibodies occur, with the same analysis for possible association with the factors listed above.

ELIGIBILITY:
Inclusion Criteria:

* Study participant who agreed to be included in the study "Studies of ongoing and completed SARS-CoV-2 infection (which causes COVID-19) within the healthcare in Stockholm County".
* Study participant who has received or will receive vaccine against Covid-19 and who gives new written consent to the study "Studies of ongoing and completed SARS-CoV-2 infection (which causes COVID-19) within the healthcare in Stockholm County, with regard to vaccinations".

Exclusion Criteria:

* those who have not given informed consent to participate in the study In this study, no initiative is taken for vaccination. The vaccinations are carried out by the healthcare system and of course follow the established exclusion and inclusion criteria for the approved vaccines. All persons who have received the vaccine and who give written consent are eligible to be included in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -Personnel within healthcare in Stockholm County who have previously participated in a study on SARS-CoV-2 infection within healthcare in Stockholm County and who are offered a vaccine against Covid-19.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 infection | 24 months post primary vaccination
  Characterized by whether they are asymptomatic infections or sick leave-requiring infections.

SECONDARY OUTCOMES:
SARS-CoV-2 antibody induction | 24 months post primary vaccination
  Antibodies will be characterized in terms of antibody levels, which SARS-CoV-2 antigen to which the response is directed and whether the antibodies are protective or not.

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Dillner, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
We have yet to determine whether the IPD will be available for other researchers.